CLINICAL TRIAL: NCT02861963
Title: Femoral Allogenic Vein Valved Conduit for Palliative Repair of Pulmonary Atresia With Ventricular Septal Defect
Brief Title: Choice of Palliative Procedures for Pulmonary Atresia With Ventricular Septal Defect Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Principal Investigator, Alexey Voitov, MD, Meshalkin Research Institute of Pathology of Circulation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FAVVC
Record Dates: First submitted 2016-07-07; First posted 2016-08-10 (Estimated); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Pulmonary Atresia With Ventricular Septal Defect; Tetralogy of Fallot With Pulmonary Atresia
Keywords: Femoral Allogenic Vein Valve Conduit; Rehabilitation of native pulmonary arteries
MeSH Terms: conditions — Pulmonary Atresia With Ventricular Septal Defect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Right ventricle outflow tract reconstruction (Experimental): RVOT reconstruction used femoral allogenic vein valve conduit through ventricular fibrillation and without VSD closure
  Interventions: Procedure: Experimental: RVOT reconstruction by femoral allogenic vein valve conduit
- Systemic-to-pulmonary artery shunts (Active Comparator): systemic-to-pulmonary artery shunts (modified Blalock-Taussig shunt)
  Interventions: Procedure: Systemic-to-pulmonary artery shunts

INTERVENTIONS:
Procedure: Experimental: RVOT reconstruction by femoral allogenic vein valve conduit — Right ventricular outflow tract reconstruction using femoral allogenic vein valve conduit under CPB and induced ventricular fibrillation
  Arms: Right ventricle outflow tract reconstruction
Procedure: Systemic-to-pulmonary artery shunts — Modified Blalock-Taussig shunt performed between the right subclavian and pulmonary arteries or the left subclavian and pulmonary arteries of the type "end to side".
  Arms: Systemic-to-pulmonary artery shunts

SUMMARY:
The aim is to compare effective growth true hypoplastic pulmonary arteries using Right Ventricle Outflow Tract Reconstruction by femoral allogenic vein valve conduit and systemic-to-pulmonary artery shunts (modified Blalock-Taussig shunt)

DETAILED DESCRIPTION:
The use of femoral allogenic vein valve conduit for Right Ventricle Outflow Tract Reconstruction is good alternative systemic-to-pulmonary artery shunts (modified Blalock-Taussig shunt). Main advantages is straight, symmetrical, pulsating, systolic blood flow in hypoplastic pulmonary artery, which stimulate growth and prepares for a radical repair. Taking into account the absence randomized studies in this area of medicine, providing investigation evaluating parameters of safety for both methodics is very actual.

ELIGIBILITY:
Inclusion criteria

Patients who met the following criteria were included:

* Patients with PA-VSD type A and B (by Tchervenkov) scheduled for palliative surgery
* Age less than one year
* Confluent pulmonary artery
* Nakata Index ≤ 120 mm2/m2. Exclusion criteria

Patients who met any of the following criteria were excluded:

* Discordant atrioventricular and/or discordant ventriculo-arterial connections
* Concomitant pathology (pneumonia, brain damage, or enterocolitis)
* Genetic syndromes (DiGeorge, Alagille, VACTER, CHARGE)
* Scheduled MAPCA unifocalisation
* Anomalous coronary arteries
* Other surgical approaches (complete primary repair, primary unification of pulmonary blood flow, stenting RVOT, or patent ductus arteriosus, radiofrequency pulmonary valve perforation).

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Growth of pulmonary arteries | From 6 to 12 months
  -Index Nakata ≥ 150 mm/m2

SECONDARY OUTCOMES:
Number of further re interventions | 1 year
  * catheterization
  * balloon plastic of the pulmonary arteries with stenting
  * unification procedures
Complications | 1 year
  * pulmonary arteries stenosis
  * Thrombosis
  * Bleeding
  * Death
  * Vein graft dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Y Omelchenko, PhD, Principal Investigator — Meshalkin Research Institute of Pathology of Circulation
Locations (1):
- Novosibirsk State Research Institute of Circulation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hibino N, He D, Yuan F, Yu JH, Jonas R. Growth of diminutive central pulmonary arteries after right ventricle to pulmonary artery homograft implantation. Ann Thorac Surg. 2014 Jun;97(6):2129-33. doi: 10.1016/j.athoracsur.2013.10.046. Epub 2014 Jan 10. PMID 24418205
- [Result] Zheng S, Yang K, Li K, Li S. Establishment of right ventricle-pulmonary artery continuity as the first-stage palliation in older infants with pulmonary atresia with ventricular septal defect may be preferable to use of an arterial shunt. Interact Cardiovasc Thorac Surg. 2014 Jul;19(1):88-94. doi: 10.1093/icvts/ivu052. Epub 2014 Mar 30. PMID 24686154
- [Result] Barozzi L, Brizard CP, Galati JC, Konstantinov IE, Bohuta L, d'Udekem Y. Side-to-side aorto-GoreTex central shunt warrants central shunt patency and pulmonary arteries growth. Ann Thorac Surg. 2011 Oct;92(4):1476-82. doi: 10.1016/j.athoracsur.2011.05.105. PMID 21958799
- [Result] Gates RN, Laks H, Johnson K. Side-to-side aorto-Gore-Tex central shunt. Ann Thorac Surg. 1998 Feb;65(2):515-6. doi: 10.1016/s0003-4975(97)01126-0. PMID 9485256
- See also: Growth of diminutive central pulmonary arteries after right ventricle to pulmonary artery homograft implantation — http://linkinghub.elsevier.com/retrieve/pii/S0003-4975(13)02368-0
- See also: Side-to-side aorto-GoreTex central shunt warrants central shunt patency and pulmonary arteries growth. — http://linkinghub.elsevier.com/retrieve/pii/S0003-4975(11)01410-X
- See also: Side-to-side aorto-Gore-Tex central shunt — http://linkinghub.elsevier.com/retrieve/pii/S0003-4975(97)01126-0